CLINICAL TRIAL: NCT01318148
Title: Prospective Trial to Evaluate Pharmacokinetic, Safety and Efficacy of Intermittent Application of Increased Doses of Caspofungin for Antifungal Prophylaxis in High Risk Patients
Brief Title: Pharmacokinetic, Safety and Efficacy of Intermittent Application of Caspofungin for Antifungal Prophylaxis
Acronym: CASPHYLAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Werner J. Heinz (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Werner J. Heinz, Consultant Infectious Diseases, Wuerzburg University Hospital
Organization: Wuerzburg University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UKW-Inf-001; 2009-015159-26 (EudraCT Number)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Fungal Infection
Keywords: Echinocandins; Caspofungin; Pharmacokinetics; Prophylaxis; Antifungal; Aspergillosis; Acute Leucemia
MeSH Terms: conditions — Mycoses; Aspergillosis | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Caspofungin (Experimental)
  Interventions: Drug: caspofungin

INTERVENTIONS:
Drug: caspofungin — Intermittent intravenous application of caspofungin
  Other Names: Cancidas

SUMMARY:
The study is a pilot phase II, prospective, non-comparative, single center trial aimed to evaluate pharmacokinetic and safety of an intermittent dosing schedule for antifungal prophylaxis in high risk patients.

DETAILED DESCRIPTION:
Pharmacokinetic and safety of caspofungin, in an intermittent dosing schedule, for prophylaxis of invasive fungal (IFI) infections will be evaluated in patients receiving induction chemotherapy for treatment of acute myeloid leukemia, myelodysplastic syndrome with blast crisis or acute lymphatic leukemia.

For prophylaxis caspofungin once daily will be given three times a week after a loading phase of three days. For drug monitoring serum samples will be collected from the first day of trial medication till one day after end of therapy (EOT). Invasive fungal infections will be diagnosed analog the criteria defined by the European organization for Research and Treatment of Cancer and the Mycosis Study Group (EORTC/MSG), revised in 2008.

Caspofungin prophylaxis will be stopped after the end of neutropenia, in case of documented proven or probable invasive fungal disease and in case of a serious adverse event attributable to the study drug, for which in view of the investigator further usage of the study drug should be avoided.

ELIGIBILITY:
Inclusion Criteria:

* acute myeloid leukemia or myelodysplastic syndrome and blast crisis or acute lymphatic leukemia
* receiving induction chemotherapy

Exclusion Criteria:

* current or need of systemic antifungal therapy
* history of proven or probable invasive aspergillus infection
* pregnant or breastfeeding women
* weight more than 100 kg
* history of allergy, hypersensitivity or any serious reaction to caspofungin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
caspofungin pharmacokinetic | day 20 (average), till end of enutropenia
  To characterize the pharmacokinetic of caspofungin IV solution in an intermittent dosing schedule of 3 times a week after a 3 days loading in a representative subject population.

SECONDARY OUTCOMES:
Caspofungin pharmacokinetic | day 20 (average), at end of neutropenia
  caspofungin serum concentrations
Incidence of invasive fungal disease and outcome | day 100 after start of chemotherapy
  Incidence of proven or probable invasive fungal disease according to the revised EORTC/MSG criteria during the period of prophylaxis and during follow up.
Safety of intermittent caspofungin | day 34 (average), 2 weeks after end of neutropenia
  Caspofungin related and all adverse and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Werner J Heinz, MD, Study Chair — University of Wuerzburg Medical Centre, Department of Internal Medicine II
Locations (1):
- University of Wuerzburg Medical Centre, Department of Internal Medicine II, Würzburg, Germany